CLINICAL TRIAL: NCT06282835
Title: The Effectiveness and Safety Study of Eravacycline Combination Therapy for Multidrug-Resistant Acinetobacter Baumannii Pneumonia
Brief Title: Eravacycline Combination Therapy for MRAB
Status: Recruiting | Type: Observational
Sponsor: Fujian Medical University Union Hospital (Other)
Responsible Party: Principal Investigator, Hui Zhang，PhD, Chief physician, Fujian Medical University Union Hospital
Other Study IDs: 2023KY242
Record Dates: First submitted 2024-01-17; First posted 2024-02-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Pulmonary Infection; Pneumonia, Bacterial; Acinetobacter Baumannii
Keywords: Eravacyline
MeSH Terms: conditions — Pneumonia, Bacterial | interventions — eravacycline

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Eravacyline combination
  Interventions: Drug: Eravacycline Injection

INTERVENTIONS:
Drug: Eravacycline Injection — Eravacycline at the recommended dose and administration method according to the instructions: 1 mg/kg intravenous administration, every 12 hours. The intravenous infusion duration is approximately 60 minutes. For patients with severe liver impairment (Child-Pugh class C), administer 1 mg/kg of this product every 12 hours on the first day, followed by 1 mg/kg every 24 hours starting from the second day.

SUMMARY:
The goal of this observational study is to learn about the eravacycline combination therapy in multidrug-resistant acinetobacter gaumannii pneumonia. The main question is to evaluate the the effectiveness and safety.

Participants will be given Eravacycline and Polymyxin，or other antibiotcs that the Investigator considered suitable. During the clinical trial, participants will be monitored for blood drug concentrations and drug concentrations in the ELF (Epithelial Lining Fluid。Clinical efficacy rate and microbiological clearance rate will be assessed at the same time

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years old;
2. Meets the diagnostic criteria for pneumonia specified by the Chinese Medical Association Respiratory Branch.
3. CRAB is identified or predominant pathogenic bacteria, and drug sensitivity test indicates that Eravacycline is sensitive to the strain;
4. Patients expected to receive Eravacycline for ≥4 days;
5. Has already signed the informed consent

Exclusion Criteria:

1. Pregnant or lactating;
2. Concurrent intracranial infection, urinary tract infection, or bloodstream infection;
3. Individuals in a moribund state;
4. The investigator believes there is any medical history, current condition, treatment, laboratory abnormalities, or other circumstances that may affect the trial results, interrupt the trial process (or the subject's inability to complete all trial requirements, operations, and visits), or increase the subject's risk with the experimental medication. Patients with terminal illnesses or evidence of immediately life-threatening diseases are excluded;
5. Patients with a history of allergic reactions to tetracyclines or any excipients in the investigational drug formulation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study plans to include patients diagnosed with CRAB pneumonia who seek medical attention at the Intensive Care Medicine Department of Fujian Medical University Union Hospital from January 2024 to April 2024
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-01-26 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical Responded Rate | 28 days
  Complete the treatment, and meet one of the following criteria to be considered clinical respond: 1. Patient's oxygenation index is stable or improved; 2. Patients with a SOFA score <3 remain unchanged or decrease, and patients with a SOFA score ≥3 decrease by at least 30%; 3. Normal body temperature for more than 3 days; 4. Improvement in pulmonary imaging; 5. Infection indicators show a continuous downward trend for 3 consecutive day

SECONDARY OUTCOMES:
The microbiological clearance rate | within 14days
  The microbiological clearance rate at the end of treatment
The all-cause mortality rate within 28 days | 28 days
  The all-cause mortality rate within 28 days
"Incidence Rate of Adverse Event | 28days
  safety data according to CTC-AE

CONTACTS AND LOCATIONS:
Overall Officials: Hui Zhang, PhD, Principal Investigator — Fujian Medical University Union Hospital
Locations (1):
- Fujian Medical University Union hospital, Fuzhou, Fujian, China